CLINICAL TRIAL: NCT04551729
Title: Fluid Restriction in Heart Failure Versus Liberal Fluid Uptake
Acronym: FRESH-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 75112
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The members of the event adjudication committee will be blinded for treatment allocation. Moreover, the statistician who performs the primary analysis will be blinded for treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid restriction (Active Comparator): Patient will receive a lifestyle advice to adhere to fluid restriction of 1500cc/day for 3 months.
  Interventions: Behavioral: Lifestyle advice for liberal fluid intake
- Liberal fluid intake (Experimental): Patient will receive a lifestyle advice for liberal fluid intake for 3 months.
  Interventions: Behavioral: Lifestyle advice for liberal fluid intake

INTERVENTIONS:
Behavioral: Lifestyle advice for liberal fluid intake — Lifestyle advice for liberal fluid intake for 3 months

SUMMARY:
Multi-centre open-label 1:1 randomized clinical trial in chronic heart failure patients on the effect of fluid restriction versus liberal fluid intake on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic HF with NYHA class II/III according to the prevailing guidelines > 6 months prior to randomization (1)
* Adult (age ≥ 18 years)

Exclusion Criteria:

* Reversible cause of HF (thyroid disorders, severe anemia, vitamin deficiencies)
* Hospital admission for HF within 3 months of randomization
* Chronic HF with NYHA class IV
* Hyponatremia at baseline (sodium <130mmol/l)
* Changes in HF medical therapy in last 14 days prior to randomization
* Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 at baseline
* Scheduled cardiac surgery within 3 months of randomization
* Recent (within 3 months) coronary intervention (PCI or CABG) or implantation of pacemaker device
* Comorbidity for which fluid restriction is advised by a different treating physician (e.g. nephrologist)
* Comorbidity with a life expectancy of less than 6 months
* The treating clinician believes that participation in the domain would not be in the best interests of the patient
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 3 months
  KCCQ Overall Summary Score (OSS) (scores minimum-maximum 0-100, higher scores indicate better outcome)

SECONDARY OUTCOMES:
Thirst distress | 3 months
  Thirst Distress Scale for patients with Heart Failure (scores minimum-maximum 8-40, higher scores indicate worse outcome)
Quality of life assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 3 months
  KCCQ Clinical Summary Score (CSS) and each of the KCCQ domains (scores minimum-maximum 0-100, higher scores indicate better outcome)
Quality of life assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 3 months
  Proportion of patients with clinically meaningful changes in KCCQ-OSS and KCCQ-CSS (improved: ≥5 points increase; stable: <5 points increase or decrease; declined: ≥5 points decrease)
Quality of life assessed with EQ-5D-5L | 3 months
  EQ-5D-5L (First part; scores minimum-maximum 0-1. Second part; (scores minimum-maximum 0-100, higher scores indicate better outcome)
Patient reported fluid intake | 6 weeks
  Patient reported fluid intake for 1 week in a fluid intake diary
Safety (Death, all-cause hospitalisations, iv loop diuretic treatment) | 6 months
  Composite of death, hospitalisations and iv loop diuretic treatment

OTHER OUTCOMES:
Safety (death, all-cause or unplanned HF hospitalisation, the requirement of iv-loop diuretics) | 6 months
  Number of occurrences of: death, all-cause or unplanned HF hospitalisation or the requirement of iv-loop diuretics
Safety (death, all-cause or unplanned HF hospitalisation, the requirement of iv-loop diuretics) | 6 months
  Time to first occurrence of: death, all-cause or unplanned HF hospitalisation or the requirement of iv-loop diuretics
Safety (acute kidney injury) | 6 months
  Number of occurrences of acute kidney injury (defined as a 50% decline in estimated glomerular filtration rate relative to baseline, or decrease of >30 ml/min/1.73m2 and to a value below 60 ml/min/1.73m2)
Safety (acute kidney injury) | 6 months
  Time to first occurrence of acute kidney injury (defined as a 50% decline in estimated glomerular filtration rate relative to baseline, or decrease of >30 ml/min/1.73m2 and to a value below 60 ml/min/1.73m2)
Serum biomarkers | 3 months
  NT-proBNP
Serum biomarkers | 3 months
  Sodium
Serum biomarkers | 3 months
  Osmolality
Serum biomarkers | 3 months
  Haemoglobin
Serum biomarkers | 3 months
  Haematocrit
Weight | 3 months
  Weight
Medication | 6 months
  Use of concomitant medication (diuretics in particular)

CONTACTS AND LOCATIONS:
Overall Officials: Roland van Kimmenade, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (8):
- Netherlands (8):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Hospital Group Twente, Almelo
  - Rijnstate Hospital, Arnhem
  - Zuyderland Ziekenhuis, Heerlen
  - Dijklander Ziekenhuis, Hoorn
  - Maastricht University Medical Centre, Maastricht
  - Bernhoven Ziekenhuis, Uden

IPD SHARING:
Plan to Share IPD: Yes
Other investigators can submit a proposal to the steering committee for the sharing of data.
  This proposal will be discussed in the steering committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Weeks
Access Criteria: These will be determined by the steering committee.

REFERENCES:
- [Background] Herrmann JJ, Beckers-Wesche F, Baltussen LEHJM, Verdijk MHI, Bellersen L, Brunner-la Rocca HP, Jaarsma T, Pisters R, Sanders-van Wijk S, Rodwell L, Van Royen N, Gommans DHF, Van Kimmenade RRJ. Fluid REStriction in Heart Failure vs Liberal Fluid UPtake: Rationale and Design of the Randomized FRESH-UP Study. J Card Fail. 2022 Oct;28(10):1522-1530. doi: 10.1016/j.cardfail.2022.05.015. Epub 2022 Jun 13. PMID 35705150
- [Result] Herrmann JJ, Brunner-La Rocca HP, Baltussen LEHJM, Beckers-Wesche F, Bekkers SCAM, Bellersen L, van Eck JWM, Hassing HC, Jaarsma T, Linssen GCM, Pisters R, Sanders-van Wijk S, Verdijk MHI, Handoko ML, van der Meer P, Verbrugge FH, Januzzi JL Jr, Bayes-Genis A, Nieuwlaat R, Rodwell L, Gommans DHF, van Kimmenade RRJ. Liberal fluid intake versus fluid restriction in chronic heart failure: a randomized clinical trial. Nat Med. 2025 Jun;31(6):2062-2068. doi: 10.1038/s41591-025-03628-4. Epub 2025 Mar 30. PMID 40159556

DOCUMENTS (6):
  • Study Protocol: Version 2.0 (First approved version) (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04551729/Prot_000.pdf
  • Study Protocol: Version 4.4 (Most recent version) (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04551729/Prot_001.pdf
  • Study Protocol: Summary of Changes V1.0 (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT04551729/Prot_002.pdf
  • Study Protocol: Summary of Changes V1.0. Appendix (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT04551729/Prot_003.pdf
  • Statistical Analysis Plan: Version 1.0 (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04551729/SAP_004.pdf
  • Statistical Analysis Plan: Version 2.0 (2024-04-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT04551729/SAP_005.pdf